CLINICAL TRIAL: NCT02689843
Title: Effects of Treatment With Cyproterone Compound-spironolactone, Metformin and Pioglitazone on Serum Inflammatory Markers in Patients With Polycystic Ovary Syndrome (PCOS)
Brief Title: Effects of Cyproterone Compound-spironolactone, Metformin and Pioglitazone on Inflammatory Markers in PCOS
Acronym: AntiPCO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of internal medicine and endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P-9145-4025
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Inflammation; Complement system proteins; Homocysteine; C-Reactive Protein; Cyproterone; Ethinyl Estradiol; Androgen Antagonists; Metformin; Thiazolidinediones; Pioglitazone
MeSH Terms: conditions — Polycystic Ovary Syndrome; Inflammation | interventions — Spironolactone; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cyproterone compound + Spironolactone (Active Comparator): Cyproterone compound (Cyproterone acetate 2mg+Ethinyl estradiol 35 mcg) once daily + Spironolactone 50 mg twice daily
  Interventions: Drug: Cyproterone compound + Spironolactone
- Metformin (Active Comparator): Metformin 1500 mg daily
  Interventions: Drug: Metformin
- Pioglitazone (Active Comparator): Pioglitazone 30 mg daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Cyproterone compound + Spironolactone — Cyproterone compound (Cyproterone Acetate 2mg-Ethinyl estradiol 35mcg) 1 tablet daily + Spironolactone 50 mg twice daily
  Other Names: CC-S
  Arms: Cyproterone compound + Spironolactone
Drug: Metformin — Metformin 500mg three times daily
  Arms: Metformin
Drug: Pioglitazone — Pioglitazone 30mg once daily
  Arms: Pioglitazone

SUMMARY:
The aim of this study is to evaluate the effects of three-month course of treatment modalities (Cyproterone compound-Spironolactone, Metformin and Pioglitazone) in patients with polycystic ovary syndrome (PCOS) on markers of inflammation [serum complement, homocysteine and high sensitive C-reactive protein (hs-CRP)] levels.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is estimated to affect up to10% of women of reproductive age, making it one of the most common endocrine disorders in this population. PCOS is associated with a broad range of adverse sequel, including hypertension, dyslipidemia, insulin resistance, hyperandrogenaemia, gestational and type 2 diabetes,which ultimately increase the cardiovascular morbidity in these patients. Also PCOS is increasingly recognized as a component of the metabolic syndrome. Management depends on symptoms or the source of androgen excess. Several treatment options are available, which allows for an individualized approach. Spironolactone is the safest potent available antiandrogen. It is effective in lowering the hirsutism score by approximately one third, although considerable individual variations exist. Other antiandrogens used to treat hirsutism and hirsutism equivalents include cyproterone acetate that has weak antiglucocorticoid effects. Metformin and thiazolidinediones, are promising adjuncts for treating PCOS. Although both of them increase insulin sensitivity, but their mechanism of action differ.

Serum complement, homocysteine and C-reactive protein (CRP) levels have been reported to be linked with insulin resistance.

The investigators want to measure serum complement, homocysteine and hs-CRP levels in patients with PCOS before and after three-month course of treatment with Cyproterone compound-Spironolactone (CC-S), metformin (M) and pioglitazone (P).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Diagnosis of Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria 2003 (two out of three required):

  1. Oligomenorrhea or anovulation
  2. Clinical and/or biochemical signs of hyperandrogenism
  3. Polycystic ovaries (by ultrasound)

Exclusion Criteria:

* Smoking
* Pregnancy
* Diabetes mellitus
* Renal failure (serum creatinine >1.5)
* Congenital adrenal hyperplasia
* Hyper or hypothyroidism
* Sex hormone therapy or antiandrogen therapy during the last three months
* Unexplained serum alanin aminotransferase (ALT) elevation more than 2.5 times above normal range
* Any systemic or febrile illnesses
* Use of glucocorticoid or anti-inflammatory drugs during the last three months
* Androgen secreting tumor
* Malignancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Serum C3 level | 3 months
  Serum concentration of a component of complement cascade: C3
Serum C4 level | 3 months
  Serum concentration of a component of complement cascade: C4
Serum high-sensitive CRP (C-reactive protein) | 3 months
  Serum concentration of high-sensitive C-reactive protein (hs-CRP)

SECONDARY OUTCOMES:
Serum total Testosterone level | 3 months
  Serum concentration of total Testosterone
Serum free Testosterone level | 3 months
  Serum concentration of free Testosterone
Serum Dehydroepiandrosterone sulfate (DHEAS) level | 3 months
  Serum concentration of Dehydroepiandrosterone sulfate
Serum follicle stimulating hormone (FSH) level | 3 months
  Serum concentration of follicle stimulating hormone
Serum luteinizing hormone (LH) level | 3 months
  Serum concentration of luteinizing hormone
Fasting Blood Sugar (FBS) | 3 months
  Fasting Blood Sugar
Fasting Serum Insulin level | 3 months
  Serum concentration of insulin
Serum homocysteine level | 3 months
  Serum concentration of homocysteine
Number of patients with adverse events | 3 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, MD, Principal Investigator — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Gholamhossein R Omrani, MD, Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No